CLINICAL TRIAL: NCT05887414
Title: Treatment Individualized Appendicitis Decision-Making (TRIAD) Patient Surveys
Brief Title: TRIAD Appendicitis Decision-making Surveys
Acronym: TRIAD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Washington (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Giana Davidson, Associate Professor: School of Medicine, University of Washington
Other Study IDs: STUDY00016171; DI-2021C3-24262 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute)
Record Dates: First submitted 2023-05-24; First posted 2023-06-02 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Appendicitis
Keywords: Decision Support Tool; Implementation; Antibiotics; Surgery
MeSH Terms: conditions — Appendicitis | interventions — BaseLine dental cement

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgery: Patients who chose to receive surgery as treatment for their appendicitis.
  Interventions: Other: Baseline; Other: 30 Day Follow Up
- Antibiotics: Patients who chose to receive antibiotics as treatment for their appendicitis.
  Interventions: Other: Baseline; Other: 30 Day Follow Up

INTERVENTIONS:
Other: Baseline — Measure Ottawa Decisional Regret at baseline when patients receive a diagnosis of appendicitis.
Other: 30 Day Follow Up — Measure Ottawa Decisional Regret after 30 days.

SUMMARY:
While appendectomy has been the main treatment of appendicitis for over 100 years, recent European studies found that, at least among highly selected patients, antibiotics alone can be an effective alternative. Surgeons and patients alike have a difficult time deciding if surgery or antibiotics are the best choice to treat appendicitis. The goal of the TRIAD is to evaluate the patients who are a part of the TRIAD implementation program and assess satisfaction and decisional regret for patients with appendicitis. This information will be used to inform the design of decision-support interventions to help patients improve their ability to make an informed decision in-line with their preferences and values.

DETAILED DESCRIPTION:
TRIAD Patient Surveys is a cross-sectional survey design that will lead to more informed decision making and better outcomes related to antibiotics for appendicitis.

TRIAD was developed from questions raised by the University of Washington CODA Trial that addressed many of the methodological issues in the European studies and included diverse, adult patients (n=1552) with almost all types of presentations of appendicitis.

TRIAD surveys will be carried out in clinics and hospitals across the United States. Patients who are diagnosed with appendicitis will be recruited for study participation regardless of which treatment (appendectomy or antibiotics) they receive. Investigators invite patients to participate in a survey designed to identify awareness of treatment options and levels of decisional conflict (measured with the Ottawa Decisional Conflict Score [DCS]). Participants will complete a baseline survey via a convenient electronic platform, and follow-up surveys will be sent at 30 days.

By implementing the TRIAD surveys, researchers hope to obtain a better understanding of patients' perspectives, knowledge, and decision-making processes regarding the choice between appendectomy and antibiotic treatment for appendicitis. This data can contribute to more informed decision-making and potentially improve outcomes related to antibiotic use for this condition.

ELIGIBILITY:
Inclusion Criteria:

* Any patient the clinical team feels is appropriate for considering either surgery or antibiotics for their initial appendicitis treatment

Exclusion Criteria:

* Pregnant patients
* Immunocompromised patients
* Patients with high complication risk of recurrent infections
* Evidence of severe phlegmon or walled off abscess or free air on imaging
* Septic shock
* Diffuse peritonitis
* Patients under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient 18+ years old or older who has been diagnosed with appendicitis at a participating TRIAD clinical site after anticipated exclusion due to age, medical condition, or radiographic finding.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Ottawa Decisional Conflict Scale | 3 years
  Ottawa Decisional Conflict Scale (DCS) measures personal perceptions of uncertainty in choosing options; modifiable factors contributing to uncertainty; and effective decision making

CONTACTS AND LOCATIONS:
Overall Officials: Giana Davidson, MD, MPH, Principal Investigator — University of Washington
Locations (17):
- United States (17):
  - Kaiser Permanente Baldwin Park, Baldwin Park, California
  - Kaiser Permanente Los Angeles, Los Angeles, California
  - Kaiser Permanente Riverside, Riverside, California
  - Grady Health System / Morehouse School of Medicine, Atlanta, Georgia
  - Northwestern Medicine, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Boston Medical Center, Boston, Massachusetts
  - Michigan Medicine- University of Michigan, Ann Arbor, Michigan
  - Columbia University Medical Center, New York, New York
  - Atrium Health, Charlotte, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Lyndon B Johnson- Harris Health, Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Texas Tech University, Lubbock, Texas
  - Harborview Medical Center, Seattle, Washington
  - Northwest Hospital and Medical Center, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington

REFERENCES:
- [Result] CODA Collaborative; Flum DR, Davidson GH, Monsell SE, Shapiro NI, Odom SR, Sanchez SE, Drake FT, Fischkoff K, Johnson J, Patton JH, Evans H, Cuschieri J, Sabbatini AK, Faine BA, Skeete DA, Liang MK, Sohn V, McGrane K, Kutcher ME, Chung B, Carter DW, Ayoung-Chee P, Chiang W, Rushing A, Steinberg S, Foster CS, Schaetzel SM, Price TP, Mandell KA, Ferrigno L, Salzberg M, DeUgarte DA, Kaji AH, Moran GJ, Saltzman D, Alam HB, Park PK, Kao LS, Thompson CM, Self WH, Yu JT, Wiebusch A, Winchell RJ, Clark S, Krishnadasan A, Fannon E, Lavallee DC, Comstock BA, Bizzell B, Heagerty PJ, Kessler LG, Talan DA. A Randomized Trial Comparing Antibiotics with Appendectomy for Appendicitis. N Engl J Med. 2020 Nov 12;383(20):1907-1919. doi: 10.1056/NEJMoa2014320. Epub 2020 Oct 5. PMID 33017106
- See also: Link to Decision Support Tool and Patient Survey — http://appyornot.org

DOCUMENTS (1):
  • Informed Consent Form (2022-08-08): https://cdn.clinicaltrials.gov/large-docs/14/NCT05887414/ICF_000.pdf